CLINICAL TRIAL: NCT03189927
Title: BD-Covered Stent for Benign Esophageal Strictures: a Safety and Feasibility Study
Acronym: BIDARCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ELLA-CS , sro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL.59222.091.16
Record Dates: First submitted 2017-05-29; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Benign Esophageal Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BD-Covered stent (Experimental): Device: BD-Covered stent for refractory benign esophageal strictures with of without fistulae
  Interventions: Device: BD-Covered esophageal stent

INTERVENTIONS:
Device: BD-Covered esophageal stent — a biodegradable covered stent is implanted to achieve a long-term relieve of dysphagia in refractory benign esophageal strictures

SUMMARY:
A non-randomized prospective clinical, pilot study in a single centre assessing the safety and feasibility of the esophageal biodegradable covered stent for refractory benign esophageal strictures with or without fistulae

DETAILED DESCRIPTION:
A non-randomized prospective clinical, pilot study in a single centre assessing the safety and feasibility of the esophageal biodegradable covered stent for refractory benign esophageal strictures with or without fistulae. The follow-up will be 6 months form implantation. After 3 months a control endoscopy will take place to evaluate stent and degradation process.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders
* Age ≥ 18 years
* Appropriate cultural level and understanding of the study
* Willingness to participate voluntarily in the study and give written informed consent
* Refractory benign esophageal stricture with or without fistulae, i.e. the patient has to pass a minimum of 2 and a maximum of 10 failed esophageal dilations to the minimal diameter of 15-mm, using a pneumatic balloon dilator or Savary bougie, not complicated by or malignancy.
* Ability to undergo periodic endoscopic follow-up.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Simultaneous participation in another clinical study
* Life expectancy of less than 12 months
* Malignant esophageal stricture
* Stenosis after laryngectomy, or if the distance between the upper edge of the stent is less than 2 cm from the upper esophageal sphincter
* Undergone an esophageal stent implantation before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment associated adverse events during follow-up (safety) | 6 months
  Short term (within 7 days after treatment) and long term (after 7 days) major complications and minor complications. Major complications are defined as life threatening and severe complications such as perforation, haemorrhage, fistula formation and severe pain. Minor complications are defined as non-life threatening or moderately severe pain and gastroesophageal reflux.
BD-Covered stent placement (feasibility): (1) ease of deployment at intended esophageal location and, (2) incidence of device related adverse events at moment of stent placement | 1 day
  Technical success is defined as ease of deployment and placement of the BD-Covered stent at the required esophageal location.

SECONDARY OUTCOMES:
Esophageal pain, measured with VAS during follow-up after stent placement | 6 months
  Pain will be measured with the VAS during follow-up
Recurrent dysphagia, measured with Ogilvie dysphagia score, during follow-up | 6 months
  Recurrent dysphagia during follow-up

IPD SHARING:
Plan to Share IPD: No